CLINICAL TRIAL: NCT01969903
Title: Effect of Dexmedetomidine Added to Lidocaine for Infra- and Supraclavicular Brachial Plexus Block
Brief Title: Study of Use of Dexmedetomidine for Regional Anesthesia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S13-00716
Record Dates: First submitted 2013-10-14; First posted 2013-10-25 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Anesthesia
Keywords: brachial plexus block; lidocaine; dexmedetomidine; bradycardia; hypotension
MeSH Terms: conditions — Bradycardia; Hypotension | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No dexmedetomidine injected (Experimental): Control group in which will be used only lidocaine for brachial plexus block
  Interventions: Drug: Precedex injection
- 0.3 microgs/kg of dexmedetomidine (Experimental): Experimental group, in which 0.3 microgs/kg dexmedetomidine will be added to lidocaine for brachial plexus block
  Interventions: Drug: Precedex injection
- 0.6 microgs/kg of dexmedeomidine (Experimental): Experimental group, in which 0.6 microgs/kg dexmedetomidine will be added to lidocaine for brachial plexus block
  Interventions: Drug: Precedex injection

INTERVENTIONS:
Drug: Precedex injection
  Other Names: precedex

SUMMARY:
The purpose of this study is to find out the proper amount of a drug called dexmedetomidine added to the local anesthetic drug called lidocaine to prolong the time and effect of pain relief provided for surgery.

Dexmedetomidine (trade name Precedex) is approved by U.S. Food and Drug Administration (FDA) and indicated for sedation (calming effect). It has both pain relieving and calming effects when added to lidocaine. In the past, addition of higher amounts of dexmedetomidine to lidocaine decreased blood pressure and heart rate. The investigators plan to study the effect of lower amounts of dexmedetomidine to achieve the same level and duration of pain relief without reduction of blood pressure and heart rate.

DETAILED DESCRIPTION:
Administered intravenously dexmedetomidine exhibits a wide range of effects that include sedation, analgesia and sympathetic activities, which translate into hemodynamic stability and anesthetic dose reduction. Recent several experimental works had demonstrated prolongation of peripheral nerve block with addition of dexmedetomidine. One human study substantiated this fact when 100µg of dexmedetomidine was added to levobupivacaine during an axillary approach brachial plexus block. This study also showed that dexmedetomidine used in this fashion resulted in lower systolic and diastolic pressures and heart rates as compared to those patients who did not receive the drug. Bradycardia requiring treatment with atropine occurred in 7 out of 30 patients (23%).

The aim of this randomized prospective study is to determine the optimal dose of dexmedetomidine added to lidocaine for infra- and supra-clavicular brachial plexus block. The investigators plan to establish a dose response relationship using 0.3µg/kg and 0.6µg/kg of dexmedetomidine added to lidocaine, epinephrine and bicarbonate mixture during infra- and supraclavicular brachial plexus block for upper extremity surgery. The doses to be used in this study are substantially lower than 100 µg dose used with levobupivacaine previously.

The investigators hypothesis is that dexmedetomidine added to lidocaine at these doses will shorten the onset and prolong the duration of brachial plexus block without significant hypotension or bradycardia.

Significant hypotension will be defined as 25% reduction of mean arterial blood pressure from the baseline or reduction of mean arterial blood pressure below 60 mm Hg.

Significant bradycardia will be defined as 25% reduction of the heart rate from the baseline or a heart rate less than 50 bpm.

ELIGIBILITY:
Inclusion Criteria:

Patients (within the age range described above) of all racial and ethnic origin, accepted to Bellevue Hospital for upper extremity surgeries, will be included in the study. Research will include only subjects who will have regional anesthesia as standard of care.

Exclusion Criteria:

The patients with history of hypersensitivity to local anesthetics, hematological diseases, bleeding or coagulation abnormalities, mental impairment, neurologic diseases, unstable cardiac, hepatic, end-stage renal, pulmonary and coagulation abnormality, history of drug abuse will not be included in the study. Vulnerable subjects also will be excluded from the study.

Patients with baseline heart rate lower than 65 bpm, blood pressure lower than 100/60, and with known allergy to precedex will be excluded from the study. Vulnerable subjects (i.e. children, pregnant women, prisoners, cognitively impaired) will be excluded from the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain scores on Visual Analog Scale will be measured | Heart rate will be monitored continuously and the blood pressure - every 5 min during the entire surgical procedure, because dexmedetomidine can cause bradycardia and hypotension. Participants will be followed for the duration of hospital stay.